CLINICAL TRIAL: NCT01282918
Title: NO Regular Defibrillation Testing In Cardioverter Defibrillator Implantation (NORDIC ICD) Trial
Brief Title: NORDIC ICD (Cardioverter Defibrillator Implantation) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NORDIC -1.1
Record Dates: First submitted 2011-01-18; First posted 2011-01-25 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Ventricular Tachyarrhythmia
Keywords: ICD; DF Test; intra-operative DF testing; VT
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Other): Patients without DF (Defibrillation) testing during ICD implantation
  Interventions: Device: ICD implantation w/o DF test
- Control group (Other): Patients with DF testing during ICD implantation (according to standardized procedure)
  Interventions: Device: ICD implantation with DF test

INTERVENTIONS:
Device: ICD implantation w/o DF test — ICD implantation without Defibrillation Test
  Arms: Study group
Device: ICD implantation with DF test — ICD implantation with DF test according to standardized procedure
  Arms: Control group

SUMMARY:
The purpose of the NORDIC ICD study is to evaluate whether ICD implantation without intra-operative DF testing is non-inferior to ICD implantation with intra-operative DF testing regarding the efficacy of the first ICD shock for the treatment of true spontaneous ventricular tachyarrhythmias.

DETAILED DESCRIPTION:
The NORDIC ICD study is justified by the need to compare the clinical outcome between patients that did receive defibrillation (DF) testing and those who did not receive DF testing during ICD implantation. The NORDIC ICD study will evaluate the impact of intra-operative DF testing on the long-term ICD first shock efficacy for true ventricular tachyarrhythmias in the observational period. Therefore, the primary analysis of this study will consider all ventricular tachyarrhythmia episodes treated by ICD shock(s) during the trial follow-up period.

Moreover, the Home MonitoringTM system of BIOTRONIK will be used in order to monitor the technical system integrity, device programming and cardiac performance continuously. It supports early information about the occurrence of VT/VF (Ventricular Tachycardia/Ventricular Fibrillation) episodes and corresponding therapies such as ICD shocks. The Home MonitoringTM capability offered by active implants has the potential to detect some of these trends early and thus to offer the possibility to intervene in time for prevention of fatal worsening of cardiac performance.

1077 patients were enrolled and randomized (1:1) in 48 centers in five European countries (Germany, Czech Republic, Denmark, Sweden and Latvia).

ELIGIBILITY:
Inclusion Criteria:

* Indication for implantation of a single chamber ICD, dual chamber ICD and CRT-D therapy according to the ACC/AHA/ESC 2006 guidelines for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death and the 2010 focused update of ESC guidelines on device therapy in heart failure (Class I recommendations)
* Primary or secondary prophylaxis
* First ICD implantation with no pre/existing or previous ICD therapy or ICD system
* The patient is willing and able to comply with the clinical investigation plan
* Patient has signed informed consent

Exclusion Criteria:

* Age ≤ 18 years
* ARVC or hypertrophic cardiomyopathy
* VF due to acute ischemia or other potentially reversible causes
* Actively listed for a transplant
* Unable or unwilling to participate in the study
* Unavailable for required follow-ups and study procedures
* Participating in another clinical study other than a registry or observational/non-interventional study
* Anticipated right sided implantation of ICD generator
* Malignant condition with a life expectancy less than the duration of the study
* Pregnant and breast-feeding women
* Terminal renal insufficiency
* Persistent AF without pre-operative TEE (Transesophageal echocardiography)
* Persistent AF with left atrial thrombus diagnosed by TEE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1077 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Average efficacy of the first ICD shock for all true ventricular tachyarrhythmias | 12 months
  The primary endpoint is the average efficacy of the first ICD shock for all true ventricular tachyarrhythmias of a patient in the observational period. More precisely, the primary endpoint will be determined as the number of true ventricular tachyarrhythmias of a patient (that were efficiently terminated by the first shock delivered by the ICD) divided by the number of true ventricular tachyarrhythmias (treated with at least one ICD shock) of the same patient.

SECONDARY OUTCOMES:
Procedural and safety endpoints | 12 months
  * Serious adverse events associated with the implantation procedure
  * Optional assessment of blood parameters indicating myocardial injury BNP (B-TYPE NATRIURETIC PEPTIDE), Creatinine, Troponin T, CK (Creatin-Kinase), CK-MB (Creatin-Kinase-MB)
  * Frequency of system revisions at implant, such as repositioning of leads, reprogramming the device to reverse polarity
  * Total fluoroscopy and implantation time
Follow-Up and efficacy endpoints | 12 months
  * All-cause mortality
  * Cardiac mortality
  * Arrhythmic mortality
  * Ventricular tachyarrhythmia conversion efficacy of the ICD shock therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Bänsch, Prof. Dr. med., Principal Investigator — Rostock University Hospital; Johan Brandt, PhD, MD, Principal Investigator — Skane University Hospital
Locations (2):
- Universitätsklinikum Rostock, Rostock, Germany
- Arrhythmia Department Skane University Hospital, Lund, Sweden

REFERENCES:
- [Background] Bansch D, Bonnemeier H, Brandt J, Bode F, Svendsen JH, Felk A, Hauser T, Wegscheider K; NORDIC ICD Trial Investigators. The NO Regular Defibrillation testing In Cardioverter Defibrillator Implantation (NORDIC ICD) trial: concept and design of a randomized, controlled trial of intra-operative defibrillation testing during de novo defibrillator implantation. Europace. 2015 Jan;17(1):142-7. doi: 10.1093/europace/euu161. Epub 2014 Aug 8. PMID 25107947